CLINICAL TRIAL: NCT01309685
Title: Effect of Varenicline on a Laboratory Model of Tobacco Addiction and on Withdrawal-Induced Cognitive Impairment
Brief Title: Effect of Varenicline on Tobacco Addiction and on Abstinence-induced Cognitive Impairment
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Purpose: Other
Other Study IDs: 999911465; 11-DA-N465
Record Dates: First submitted 2011-03-04; First posted 2011-03-07 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2012-11-26

CONDITIONS: Drug Addiction
Keywords: Cognition; Smoking; Nicotine; Varenicline; Withdrawal
MeSH Terms: conditions — Substance-Related Disorders; Smoking | interventions — Varenicline

INTERVENTIONS:
Drug: Varenicline

SUMMARY:
Background:

- Varenicline (Chantix ) is a drug that is approved by the Food and Drug Administration (FDA) to help people stop smoking. Varenicline is very effective in helping some people quit smoking, but is less effective for others. Researchers are interested in conducting more in-depth studies into how varenicline works, including its effect on smokers' responses to items that may trigger cigarette cravings, in order to develop better smoking cessation medications.

Objectives:

- To examine the effectiveness of varenicline as an effective medication for tobacco addiction by studying its effect on nicotine reinforcement, nicotine-seeking behavior, cue-elicited craving, and performance impairment and craving after overnight tobacco deprivation.

Eligibility:

- Individuals between 18 and 50 years of age who have been smoking at least 10 cigarettes per day for at least 2 years.

Design:

* This study will require 12 study visits. Some visits will be brief and other visits that involve test sessions will last up to 8 hours. If no sessions are repeated, the study will take 26 days. Participants will not be required to attempt to quit smoking during this study.
* Participants will be screened with a full physical examination and medical history, blood and urine tests, and other tests as required by the study researchers.
* Participants will take two sets of pills during the study: the first set during the first 12 days of the study, followed by a 2-day break, then the second set during the last 12 days. Some of the pills will contain varenicline, and others will be placebos.
* On Day 1 of the study, participants will come to the National Institute on Drug Abuse to receive the first set of pills. Participants will take the first pill before leaving.
* On Day 8, participants will have a training session that will measure the amount of carbon monoxide in the breath. Participants will also complete several questionnaires about smoking habits and current mood, and will have a chance to practice the procedures they will do in the study.
* On Days 9 and 10, participants will have behavioral test sessions that will last 7 to 8 hours. Day 9 will involve tests of cue response to items that may trigger cigarette cravings, and tests of general nicotine cravings over several hours. Day 10 will involve tests of general nicotine cravings over several hours, and then tests of nicotine-seeking behavior. Participants will be provided with lunch during these all-day sessions.
* On Day 11, participants will have memory and attention tests, and will provide a blood sample. Participants will not be allowed to smoke for 12 hours before the start of the next test on Day 12.
* On Day 12, participants will provide a breath sample, and will have two sets of memory and attention tests before they will be permitted to start smoking again. There will be no tests on Days 13 and 14.
* Starting on Day 15, participants will repeat the schedule of tests from Days 1 through 12 with the second set of pills.

DETAILED DESCRIPTION:
Objectives

1. To examine several potential mechanisms by which varenicline functions as an effective medication for tobacco addiction: a) nicotine reinforcement (forced-choice procedure), b) nicotine-seeking behavior (operant response task), c) cue-elicited craving, and d) performance impairment and craving after overnight tobacco deprivation.
2. To validate our laboratory measures by using a medication with known efficacy in the treatment of tobacco addiction.

Study population

The study will enroll 50 healthy adult smokers to attain 25 completers.

Design

The study is a placebo-controlled, crossover design comparing the effects of varenicline and placebo.

Outcome Measures

During cue-reactivity sessions, primary measures include tobacco craving, mood, and autonomic responsivity (heart rate, blood pressure, skin conductance, and skin temperature). During forced-choice sessions, the primary measure is the percentage of nicotine cigarette puffs chosen during choice trials. During operant response sessions, primary measures include breakpoint (final ratio completed), total number of responses, and number of cigarette puffs earned and taken. During the tobacco deprivation session, primary measures include self-reported withdrawal, tobacco craving, mood, and cognitive task performance (accuracy and response time).

Secondary study measures include baseline demographic and smoking history, level of nicotine dependence, tobacco craving, and mood.

ELIGIBILITY:
* INCLUSION CRITERIA:
* 18-50 year old males and females
* smoking at least 10 cigarettes per day for at least 2 years
* estimated IQ score greater than or equal to 85
* medically and psychologically healthy as determined by screening criteria

EXCLUSION CRITERIA:

* definite plan to reduce or quit tobacco use in the next 30 days
* treatment for tobacco dependence in the past 3 months
* use of nicotine replacement products, bupropion, or varenicline in the past 3 months as an aid to quit or reduce smoking
* use of any oral tobacco product in the past 6 months
* history of drug or alcohol dependence within last 5 years
* consumption of more than 15 alcoholic drinks per week on average during the past month
* use of any illicit drug more than once per week on average during the past month
* current use of any medication that would interfere with the protocol in the opinion of MAI
* pregnant, nursing, or become pregnant during the study
* HIV positive

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-02-13; Primary Completion 2014-11-26 (Actual); Study Completion 2014-11-26 (Actual)

PRIMARY OUTCOMES:
Tobacco craving, nicotine reinforcement, cognitive performance

SECONDARY OUTCOMES:
Nicotine dependence, smoking history, mood

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Heishman, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)

REFERENCES:
- [Background] Bell SL, Taylor RC, Singleton EG, Henningfield JE, Heishman SJ. Smoking after nicotine deprivation enhances cognitive performance and decreases tobacco craving in drug abusers. Nicotine Tob Res. 1999 Mar;1(1):45-52. doi: 10.1080/14622299050011141. PMID 11072387
- [Background] Bickel WK, Hughes JR, DeGrandpre RJ, Higgins ST, Rizzuto P. Behavioral economics of drug self-administration. IV. The effects of response requirement on the consumption of and interaction between concurrently available coffee and cigarettes. Psychopharmacology (Berl). 1992;107(2-3):211-6. doi: 10.1007/BF02245139. PMID 1615122
- [Background] Burstein AH, Fullerton T, Clark DJ, Faessel HM. Pharmacokinetics, safety, and tolerability after single and multiple oral doses of varenicline in elderly smokers. J Clin Pharmacol. 2006 Nov;46(11):1234-40. doi: 10.1177/0091270006291837. PMID 17050788